CLINICAL TRIAL: NCT05311358
Title: The Engineer-Built System, Video-Game Based Kinect Sensor in Upper Extremities Problems in Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Warakorn Charoensuk (Unknown); Apiphan Iamchaimongkol (Unknown); Tulyapruek Tawonsawatruk (Unknown)
Responsible Party: Principal Investigator, Sivaporn Vongpipatana, Assistant Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MURA2021/768
Record Dates: First submitted 2022-03-08; First posted 2022-04-05 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
Keywords: video-game based Kinect sensor; upper extremities
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: In the first phase, we will test our video-game based Kinect sensor in healthy children aged 10-12 years old. The healthy children and the occupational therapists have to reply the satisfaction form and comment our game for further improvement. The sample size of this phase is 10.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal children (Experimental): Normal children aged 10-15 years play the game and comment on the satisfaction form
  Interventions: Device: The engineer-built system, video-game based Kinect sensor

INTERVENTIONS:
Device: The engineer-built system, video-game based Kinect sensor — There are 3 computer games using Kinect sensor to detect movement of trunk and upper extremities of the children.

SUMMARY:
There are 3 phases of this project. First phase is to study the satisfaction in healthy children aged 10-15 years old when they are playing our computer games. The sample size of this phase was 10. In addition, we will ask the occupational therapist to play and comment our game for further development.

ELIGIBILITY:
Inclusion Criteria:

* Normal children aged 10-15 years
* Sufficient cognitive/attention capacity
* Give the informed consent

Exclusion Criteria:

* Inability to understand the instruction and follow the task
* Has severe visual or auditory impairment
* Has limb deformities that interfere with video game playing
* Got an epilepsy or convulsive condition
* Denied to give the informed consent

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
satisfaction form | immediately after playing game
  The satisfaction form will be evaluated by healthy children. The satisfaction form will ask the children to rate the games in the following subjects: the presentation of game, the contents of game, the convenience for users the feeling after playing and the further suggestion about the games. There are 5-likert-scale in the satisfaction form: totally disagree, disagree, neutral, agree and totally agree.

SECONDARY OUTCOMES:
Satisfaction form | immediately after playing game
  The satisfaction form will be evaluated by occupational therapists. The satisfaction form will ask the therapist to rate the games in the following subjects: the presentation of game, the contents of game, the convenience for users the feeling after playing and the further suggestion about the games. There are 5-likert-scale in the satisfaction form: totally disagree, disagree, neutral, agree and totally agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
I will share the information on satisfaction form with the engineers who developed game for game improvement.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol will be share among the researcher team during study period. The statistical analysis plan will be share with the statistician during the analysis and summarize period.
Access Criteria: using code number of the participants

REFERENCES:
- [Background] Arneson CL, Durkin MS, Benedict RE, Kirby RS, Yeargin-Allsopp M, Van Naarden Braun K, Doernberg NS. Prevalence of cerebral palsy: Autism and Developmental Disabilities Monitoring Network, three sites, United States, 2004. Disabil Health J. 2009 Jan;2(1):45-8. doi: 10.1016/j.dhjo.2008.08.001. PMID 21122742
- [Background] Bhasin TK, Brocksen S, Avchen RN, Van Naarden Braun K. Prevalence of four developmental disabilities among children aged 8 years--Metropolitan Atlanta Developmental Disabilities Surveillance Program, 1996 and 2000. MMWR Surveill Summ. 2006 Jan 27;55(1):1-9. PMID 16437058
- [Background] Paneth N, Hong T, Korzeniewski S. The descriptive epidemiology of cerebral palsy. Clin Perinatol. 2006 Jun;33(2):251-67. doi: 10.1016/j.clp.2006.03.011. PMID 16765723
- [Background] Prevalence and characteristics of children with cerebral palsy in Europe. Dev Med Child Neurol. 2002 Sep;44(9):633-40. PMID 12227618
- [Background] Chen YP, Lee SY, Howard AM. Effect of virtual reality on upper extremity function in children with cerebral palsy: a meta-analysis. Pediatr Phys Ther. 2014 Fall;26(3):289-300. doi: 10.1097/PEP.0000000000000046. PMID 24819682
- [Background] 7. Samia Abdel Rahman, Abdel Rahman, Afaf A. Shaheen. Virtual Reality Use in Motor Rehabilitation of Neurological Disorders: A Systematic Review. Middle-East Journal of Scientific Research; 7 (1): 63-70.
- [Background] Chen YP, Kang LJ, Chuang TY, Doong JL, Lee SJ, Tsai MW, Jeng SF, Sung WH. Use of virtual reality to improve upper-extremity control in children with cerebral palsy: a single-subject design. Phys Ther. 2007 Nov;87(11):1441-57. doi: 10.2522/ptj.20060062. Epub 2007 Sep 25. PMID 17895352
- [Background] Green D, Wilson PH. Use of virtual reality in rehabilitation of movement in children with hemiplegia--a multiple case study evaluation. Disabil Rehabil. 2012;34(7):593-604. doi: 10.3109/09638288.2011.613520. Epub 2011 Oct 6. PMID 21978233
- [Background] Pruksananonda C. Cerebral palsy. In: Prasongjean P, editor. Cerebral Palsy. Bangkok: Chulolongkorn University Printing House; 2010. p. 1-3.